CLINICAL TRIAL: NCT01987102
Title: An Open-Label, Multicenter, Phase I/II Clinical Trial to Identify the Modufolin® Dose With Most Favorable Safety Prospect and Confirmed Ability to Mitigate High-Dose Methotrexate Induced Toxicity During Treatment of Osteosarcoma Patients
Brief Title: Investigation of [6R] 5,10-methylenetetrahydrofolate (Arfolitixorin) as Rescue Therapy for Osteosarcoma Patients Treated With HDMTX.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Isofol Medical AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ISO-MTX-003
Record Dates: First submitted 2013-11-05; First posted 2013-11-19 (Estimated); Results first posted 2019-06-26 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Osteosarcoma
Keywords: Methotrexate; Rescue treatment
MeSH Terms: conditions — Osteosarcoma | interventions — Leucovorin; 5,10-methylenetetrahydrofolic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): 1 MAP cycle (incl. 2 HDMTX Courses using Calcium Folinate rescue 15mg/m2)
  1 MAP cycle (incl. 2 HDMTX Courses using [6R] 5,10-methylenetetrahydrofolate rescue 15mg/m2)
  Interventions: Drug: Calcium Folinate; Drug: [6R] 5,10-methylenetetrahydrofolate (arfolitixorin)
- Cohort 2 (Experimental): 1 MAP cycle (incl. 2 HDMTX Courses using Calcium Folinate rescue 15mg/m2)
  1 MAP cycle (incl. 2 HDMTX Courses using [6R] 5,10-methylenetetrahydrofolate rescue 7,5mg/m2 or 30mg/m2*)
  *Dose will depend on outcome from Cohort 1
  Interventions: Drug: Calcium Folinate; Drug: [6R] 5,10-methylenetetrahydrofolate (arfolitixorin)

INTERVENTIONS:
Drug: Calcium Folinate — The enrolled patients will be treated according to the MAP schedule and will receive the study drug Calcium Folinate commencing 24 hours after the administration of HDMTX and then every 6 hours (q6h) thereafter until the S-MTX levels are ≤ 0.1 µmol/L, in accordance with COG management recommendations.
  All patients will receive standard o care (SOC) in the two (2) first HDMTX courses and [6R] 5,10-methylenetetrahydrofolate in the two (2) following courses. Patients will be enrolled in two (2) [6R] 5,10-methylenetetrahydrofolate dose cohort groups: with [6R] 5,10-methylenetetrahydrofolate start dose of 15 mg/m2 (i.e. the same as for SOC rescue) the first cohort will be administered, and 7.5 or 30 mg/m2 in the second cohort.
  Other Names: Leucovorin
Drug: [6R] 5,10-methylenetetrahydrofolate (arfolitixorin) — The enrolled patients will be treated according to the MAP schedule and will receive the study drug [6R] 5,10-methylenetetrahydrofolate commencing 24 hours after the administration of HDMTX and then every 6 hours (q6h) thereafter until the S-MTX levels are ≤ 0.1 µmol/L, in accordance with COG management recommendations.
  All patients will receive standard o care (SOC) in the two (2) first HDMTX courses and [6R] 5,10-methylenetetrahydrofolate in the two (2) following courses. Patients will be enrolled in two (2) [6R] 5,10-methylenetetrahydrofolate® dose cohort groups: with [6R] 5,10-methylenetetrahydrofolate start dose of 15 mg/m2 (i.e. the same as for SOC rescue) the first cohort will be administered, and 7.5 or 30 mg/m2 in the second cohort.
  Other Names: Modufolin; arfolitixorin

SUMMARY:
An open-label, multicenter, phase I/II clinical trial to identify the [6R] 5,10-methylenetetrahydrofolate (arfolitixorin) dose with most favorable safety prospect and confirmed ability to mitigate high-dose methotrexate induced toxicity during treatment of osteosarcoma patients

DETAILED DESCRIPTION:
This is a non-blinded, multicenter, exploratory study in osteosarcoma patients. The study focuses on the overall safety of the HDMTX courses given within a Methotrexate, Adriamycin (doxorubin) and cisPlatin (MAP) treatment schedule, which is closely related to the efficacy of the concomitantly administered folate rescue treatment. Additionally the study aimes to collect pharmacokinetic (PK) profiles of metotrexate (MTX) in serum, of folate metabolites in plasma and to decide the Modufolin® dose to use in future studies.

Patients are enrolled in the study at the first, third or the fifth HDMTX course in a MAP treatment schedule and receive folate rescue therapy according to a strategy based on the Children's Oncology Group (COG) treatment management recommendations used in study protocol AOST0331.

Folate rescue treatment with Calcium Folinate (SOC) or Modufolin® (MOD) commence 24 h after start of HDMTX administration and then every 6 h until the serum MTX levels are ≤0.1 μmol/L. In case delayed MTX elimination occurs with significant increase in S-creatinine and/or occurrence of oral mucositis or signs of hypo cellular bone marrow, the folate rescue dose and/or the administered hydration will be adjusted in accordance with the COG based MTX toxicity management recommendations.

All patients receives SOC (15 mg/m2) in the first 2 HDMTX courses and MOD in the following 2 courses. Patients are enrolled in one of two MOD dose cohorts: Cohort 1 (15 mg/m2) and Cohort 2 (30 or 7.5 mg/m2 depending on outcome of Cohort 1). Only patients with successful advancements from the first 2 HDMTX courses with Calcium Folinate are allowed to continue with MOD as rescue in the following MAP cycle.

Safety data will be reviewed by an independent board, Data and Safety Monitoring Board (DSMB) that will assess each patient and made recommendations regarding the enrolment of subsequent patients. Furthermore, the DSMB will make a dose level recommendation for Cohort 2 and also a recommendation whether younger children may be allowed in this cohort.

ELIGIBILITY:
Main Inclusion Criteria (HDMTX with SOC rescue):

* Patients must have histological evidence of osteosarcoma (metastatic disease accepted).
* Patients must be eligible for HDMTX according to the MAP treatment schedule described in the study protocol and fulfill all of the criteria below prior to first course of HDMTX in the study.

  1. Serum MTX: ≤0.1μmol/L
  2. Neutrophils: ≥0.25x109/L
  3. Platelets: ≥50x109/L
  4. Serum bilirubin: ≤1.25x upper limit of normal (ULN)
  5. Glomerular filtration rate (GFR) ≥70 mL/min/1.73m2
  6. No adverse event (AE) Grade 2 or more (NCI CTCAE v4.0) related to HDMTX hindering a potential HDMTX administration, at the discretion of the investigator.
* Patients must be 12-40 years of age. This age range may be extended with younger patients for enrolment in Cohort 2 if collected data from Cohort 1 support this and it is recommended by the DSMB.

Exclusion criteria for enrolment:

* Involvement in another clinical trial within 30 days before enrolment in the study.
* Hypersensitivity to Calcium Folinate.
* Previous treatment with glucarpidase.
* Known serious concomitant systemic disorders (e.g., active infection including HIV, liver dysfunction, cardiac disease) that, in the opinion of the investigator, would compromise the patient's ability to complete the study

Main Inclusion criteria for continuation (HDMTX treatment with Modufolin rescue):

* Patients, who were included in the study in accordance with the inclusion criteria above, must have received 2 adjacent courses of HDMTX with SOC rescue according to the MAP treatment schedule in accordance with this study protocol.
* Patients eligible for continued HDMTX according to the MAP treatment schedule and with a history of successful advancement from first to second HDMTX course within the previous MAP cycle
* Patients eligible for continued HDMTX according to the MAP treatment schedule and with a history of successful advancement to next MAP cycle after end of previous MAP cycle
* No significant changes to the patient's medical condition from the start of the study that in the opinion of the investigator would compromise the patient's ability to complete the study.
* Patients who have undergone surgical resection of their tumor must have recovered from their surgery and be eligible to continue on the MAP regimen; any post-operative complications should be resolved to NCI CTCAE v4.0 Grade 1 or better.

Ages: 6 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-01-03 (Actual); Study Completion 2017-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Eriksson, MD PhD, Principal Investigator — Department of Oncology, Skåne University Hospital
Locations (5):
- Czechia (2):
  - Fakultní nemocnice Brno Klinika detske onkologie, Brno
  - Fakultní nemocnice v Motole, Prague
- Semmelweis Egyetem II. Sz. Gyermekgyógyászati Klinika, Budapest, Hungary
- Instytut Matki i Dziecka, Warsaw, Poland
- Department of Oncology, Skåne University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were pre-screened for eligibility to participate by the principal investigator among those patients who have received confirmed diagnosis of osteosarcoma and were planned for surgical resection of their tumor in combination with neoadjuvant or adjuvant chemotherapy.
Groups:
- Cohort 1: 1 MAP cycle (incl. 2 HDMTX courses with Calcium Folinate (SOC) rescue 15mg/m2)
  1 MAP cycle (incl. 2 HDMTX courses with Modufolin (MOD) rescue 15mg/m2)
  Treatment according to the MAP schedule applied. SOC or MOD commenced 24 h after administration of HDMTX and then every 6 h until the serum-MTX levels were ≤ 0.1 µmol/L, in accordance with COG management recommendations.
- Cohort 2: 1 MAP cycle (incl. 2 HDMTX courses with Calcium Folinate (SOC) rescue 15mg/m2)
  1 MAP cycle (incl. 2 HDMTX courses with Modufolin (MOD) rescue 7.5mg/m2)
  Treatment according to the MAP schedule applied. SOC or MOD commenced 24 h after administration of HDMTX and then every 6 h until the serum-MTX levels were ≤ 0.1 µmol/L, in accordance with COG management recommendations.
Period: 2 Courses of HDMTX With SOC Rescue
Arm/Group | Cohort 1 | Cohort 2
Started | 8 | 10
Completed | 4 | 4
Not Completed | 4 | 6
Not completed — Adverse Event | 2 | 2
Not completed — Laboratory abnormality | 1 | 2
Not completed — Change in planned chemotherapy | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Incorrectly included | 0 | 1
Period: 2 Courses of HDMTX With MOD Rescue
Arm/Group | Cohort 1 | Cohort 2
Started | 4 | 4
Completed | 4 | 3
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 8 | 10 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 8 | 16
  Between 18 and 65 years | 0 | 2 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 7 | 8 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 10 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Sweden | 0 | 1 | 1
  Hungary | 2 | 1 | 3
  Czechia | 5 | 6 | 11
  Poland | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of AEs Per Severity (All Courses)
Description: Characterization (number and severity grade) of toxicity reported for each course of HDMTX treatment with folate rescue therapy and continuing until eight (8) days after start of HDMTX administration, per NCI CTCAE v4.0 (Grade refers to the severity of the AE). The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE; Grade 1 Mild, Grade 2 Moderate, Grade 3 Severe, Grade 4 Life-threatening, and Grade 5 Death related to AE.
Time Frame: From the start of HDMTX administration through 8 days post dose for each course of HDMTX in total
Population: The All Patients Treated Set (APTS) included all patients receiving at least one bolus injection of Modufolin (MOD).
Measure: Number; unit: Number of AEs
Groups:
- Cohort 2: 1 MAP cycle (incl. 2 HDMTX courses with SOC rescue 15mg/m2)
  1 MAP cycle (incl. 2 HDMTX courses with MOD rescue 7.5mg/m2)
  Treatment according to the MAP schedule applied. SOC or MOD commenced 24 h after administration of HDMTX and then every 6 h until the serum-MTX levels were ≤ 0.1 µmol/L, in accordance with COG management recommendations.
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 4 | 4
Number of AEs
  Grade 1 | 40 | 27
  Grade 2 | 8 | 15
  Grade 3 | 11 | 6
  Grade 4 | 3 | 1

2. Primary Outcome: Number of HDMTX Related AEs Per Severity (All Courses)
Description: Characterization (frequency and severity grade) of toxicity reported for each course of HDMTX treatment with folate rescue therapy and continuing until eight (8) days after start of HDMTX administration, per NCI CTCAE v4.0 (Grade refers to the severity of the AE). The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE; Grade 1 Mild, Grade 2 Moderate, Grade 3 Severe, Grade 4 Life-threatening, and Grade 5 Death related to AE.
Time Frame: From the start of HDMTX administration through 8 days post dose for each course of HDMTX in total
Population: The All Patients Treated Set (APTS) included all patients receiving at least one bolus injection of Modufolin (MOD).
Measure: Number; unit: Number of AEs
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 4 | 4
Number of AEs
  Grade 1 | 25 | 20
  Grade 2 | 6 | 12
  Grade 3 | 6 | 5
  Grade 4 | 1 | 1

3. Primary Outcome: Number of Ongoing AEs Per HDMTX Course
Description: as for outcome 2
Time Frame: From the start of HDMTX administration through 8 days post dose for each course of HDMTX
Population: The All Patients Treated Set (APTS) included all patients receiving at least one bolus injection of Modufolin (MOD).
Measure: Number; unit: Number of AEs
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 4 | 4
Number of AEs
  Course 1 (SOC) | 14 | 10
  Course 2 (SOC) | 19 | 10
  Course 1 (MOD) | 6 | 10
  Course 2 (MOD) | 14 | 16

4. Primary Outcome: Number of Ongoing HDMTX Related AEs Per HDMTX Course
Description: as for outcome 2
Time Frame: From the start of HDMTX administration through 8 days post dose for each course of HDMTX
Population: The All Patients Treated Set (APTS) included all patients receiving at least one bolus injection of Modufolin (MOD).
Measure: Number; unit: Number of AEs
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 4 | 4
Number of AEs
  Course 1 (SOC) | 13 | 8
  Course 2 (SOC) | 13 | 8
  Course 1 (MOD) | 5 | 10
  Course 2 (MOD) | 12 | 16

5. Secondary Outcome: Number of Administered HDMTX Courses Classified as Having Met the Criteria for Successful Advancement According to Definition A and/or Definition B
Description: Definition A: Successful advancement from 1st to 2nd HDMTX course within the same MAP cycle. Fulfilling all of the following criteria 8 days after start of first HDMTX course within the same MAP cycle:
  1. Serum MTX: ≤0.1μmol/L
  2. Neutrophils: ≥0.25x109/L
  3. Platelets: ≥50x109/L
  4. Serum bilirubin: ≤1.25 x upper limit of normal (ULN)
  5. Glomerular filtration rate (GFR) ≥70 mL/min/1.73m2
  6. No AE Grade 2 or more related to HDMTX hindering a potential HDMTX administration, at the discretion of the investigator
  Definition B: Successful advancement to next MAP cycle
  Fulfilling all of the following criteria 8 days after start of the second HDMTX course in previous MAP cycle:
  1. Serum MTX: ≤0.1μmol/L
  2. Neutrophils: ≥ 0.75 x 109/L
  3. Platelets: ≥75x109/L
  4. Serum bilirubin: ≤1.25xULN
  5. GFR ≥70 mL/min/1.73m2
  6. No AE Grade 2 or more related to HDMTX hindering a potential Adriamycin/Doxorubicin and Cisplatin (AP) administration, at the discretion of the investigator
Time Frame: 8 days after start of first and/or second HDMTX course in a MAP cycle
Population: The All Patients Treated Set (APTS) included all patients receiving at least one bolus injection of Modufolin (MOD).
Measure: Number; unit: Number of courses
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 4 | 4
Number of courses
  Successful Course SOC 1 | 4 | 4
  Unsuccessful Course SOC 1 | 0 | 0
  Successful Course SOC 2 | 4 | 4
  Unsuccessful Course SOC 2 | 0 | 0
  Successful Course MOD 1 | 4 | 3
  Unsuccessful Course MOD 1 | 0 | 1
  Successful Course MOD 2 | 4 | 2
  Unsuccessful Course MOD 2 | 0 | 1

6. Secondary Outcome: Number of Administered MAP Cycles Classified as Having Met the Criteria for Successful Advancement From First to Second HDMTX Course Within the Same MAP Cycle According to Definition A.
Description: Definition A: Successful advancement from first to second HDMTX course within the same MAP cycle
  Fulfilling all of the following criteria 8 days after start of first HDMTX course within the same MAP cycle:
  1. Serum MTX: ≤ 0.1 μmol/L
  2. Neutrophils: ≥ 0.25 x 109/L
  3. Platelets: ≥ 50 x 109/L
  4. Serum bilirubin: ≤ 1.25 x ULN
  5. GFR ≥ 70 mL/min/1.73 m2
  6. No AE Grade 2 or more (NCI CTCAE v4.0) related to HDMTX hindering a potential HDMTX administration, at the discretion of the investigator
Time Frame: 8 days after start of first HDMTX course in a MAP cycle
Population: The All Patients Treated Set (APTS) included all patients receiving at least one bolus injection of Modufolin (MOD).
Measure: Number; unit: Number of courses
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 4 | 4
Number of courses
  Successful Course SOC 1 | 4 | 4
  Unsuccessful Course SOC 1 | 0 | 0
  Successful Course MOD 1 | 4 | 3
  Unsuccessful Course MOD 1 | 0 | 1

7. Secondary Outcome: Number of Administered MAP Cycles Classified as Having Met the Criteria for Successful Advancement to Next MAP Cycle According to Definition B.
Description: Definition B: Successful advancement to next MAP cycle
  Fulfilling all of the following criteria 8 days after start of the second HDMTX course in previous MAP cycle:
  1. Serum MTX: ≤ 0.1 μmol/L
  2. Neutrophils: ≥ 0.75 x 109/L
  3. Platelets: ≥ 75 x 109/L
  4. Serum bilirubin: ≤ 1.25 x ULN
  5. GFR ≥ 70 mL/min/1.73 m2
  6. No AE Grade 2 or more (NCI CTCAE v4.0) related to HDMTX hindering a potential Adriamycin/Doxorubicin and Cisplatin (AP) administration, at the discretion of the investigator
Time Frame: 8 days after start of second HDMTX course in a MAP cycle
Population: The All Patients Treated Set (APTS) included all patients receiving at least one bolus injection of Modufolin (MOD).
Measure: Number; unit: Number of courses
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 4 | 4
Number of courses
  Successful Course SOC 2 | 4 | 4
  Unsuccessful Course SOC 2 | 0 | 0
  Successful Course MOD 2 | 4 | 2
  Unsuccessful Course MOD 2 | 0 | 1

8. Secondary Outcome: Time to Successful MTX Elimination (Definition C)
Description: Definition C: Time to successful MTX elimination = Time from start of MTX treatment until serum MTX level is ≤ 0.1 μmol/L
Time Frame: Time from start of MTX treatment until serum MTX level is ≤ 0.1 μmol/L
Population: The All Patients Treated Set (APTS) included all patients receiving at least one bolus injection of Modufolin (MOD).
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 4 | 4
hours
  Time (h) Course SOC 1 | 84.52 (15.00) | 62.75 (3.21)
  Time (h) Course SOC 2 | 77.0 (19.60) | 62.75 (9.91)
  Time (h) Course MOD 1 | 74.00 (15.87) | 65.75 (11.50)
  Time (h) Course MOD 2 | 72.50 (15.78) | 88.0 (43.41)

9. Secondary Outcome: Number of HDMTX Courses in Which the Initial Hydration Was Increased
Time Frame: Time from start of MTX treatment until serum MTX level is ≤ 0.1 μmol/L
Population: The All Patients Treated Set (APTS) included all patients receiving at least one bolus injection of Modufolin (MOD).
Measure: Number; unit: HDMTX courses
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 4 | 4
HDMTX courses
  Hydration change in Course SOC 1 | 2 | 0
  Unchanged hydration Course SOC 1 | 2 | 4
  Hydration change in Course SOC 2 | 1 | 0
  Unchanged hydration Course SOC 2 | 3 | 4
  Hydration change in Course MOD 1 | 2 | 2
  Unchanged hydration Course MOD 1 | 2 | 2
  Hydration change in course MOD 2 | 2 | 1
  Unchanged hydration Course MOD 2 | 2 | 2

10. Secondary Outcome: Number of HDMTX Courses With Delayed MTX Elimination (Definition D).
Description: Definition D: Delayed MTX elimination (according to COGs excretion toxicity management instructions)
  S-MTX levels of:
  > 10 μmol/L at 24 h after start of MTX administration, OR > 1 μmol/L at 48 h after start of MTX administration, OR > 0.1 μmol/L at 72 h after start of MTX administration or later
Time Frame: Time from start of MTX treatment until serum MTX level is ≤ 0.1 μmol/L
Population: The All Patients Treated Set (APTS) included all patients receiving at least one bolus injection of Modufolin (MOD).
Measure: Number; unit: Number of courses
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 4 | 4
Number of courses
  Delayed MTX elimination in Course SOC 1 | 3 | 0
  Undelayed MTX elimination in Course SOC 1 | 1 | 4
  Delayed MTX elimination in Course SOC 2 | 3 | 1
  Undelayed MTX elimination in Course SOC 2 | 1 | 3
  Delayed MTX elimination in Course MOD 1 | 2 | 1
  Undelayed MTX elimination in Course MOD 1 | 2 | 3
  Delayed MTX elimination in Course MOD 2 | 2 | 1
  Undelayed MTX elimination in Course MOD 2 | 2 | 2

11. Secondary Outcome: Number of HDMTX Courses With Delayed Early MTX Elimination (Definition E).
Description: Definition E: Delayed early MTX elimination (according to US label for Calcium Folinate)
  S-MTX levels of:
  * 50 μmol/L at 24 hours after start of MTX administration, OR
  * 5 μmol/L at 48 hours after start of MTX administration OR An increase in S-Creatinine level of 100% or greater at 24 hours after start of MTX administration.
Time Frame: Time from start of MTX treatment until serum MTX level is ≤ 0.1 μmol/L
Population: The All Patients Treated Set (APTS) included all patients receiving at least one bolus injection of Modufolin (MOD).
Measure: Number; unit: Number of courses
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 4 | 4
Number of courses
  Delayed early MTX elimination in Course SOC 1 | 0 | 0
  Undelayed early MTX elimination in Course SOC 1 | 4 | 4
  Delayed early MTX elimination in Course SOC 2 | 0 | 0
  Undelayed early MTX elimination in Course SOC 2 | 4 | 4
  Delayed early MTX elimination in Course MOD 1 | 0 | 0
  Undelayed early MTX elimination in Course MOD 1 | 4 | 4
  Delayed early MTX elimination in Course MOD 2 | 0 | 0
  Undelayed early MTX elimination in Course MOD 2 | 4 | 3

12. Secondary Outcome: Number of HDMTX Courses With Delayed Late MTX Elimination (Definition F).
Description: Definition F: Delayed late MTX elimination (according to US label for Calcium Folinate)
  S-MTX level:
  > 0.2 μmol/L at 72 hours AND > 0.1 μmol/L at 96 hours after start of MTX administration.
Time Frame: Time from start of MTX treatment until serum MTX level is ≤ 0.1 μmol/L
Population: The All Patients Treated Set (APTS) included all patients receiving at least one bolus injection of Modufolin (MOD).
Measure: Number; unit: Number of courses
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 4 | 4
Number of courses
  Delayed late MTX elimination in Course SOC 1 | 0 | 0
  Undelayed late MTX elimination in Course SOC 1 | 3 | 1
  Delayed late MTX elimination in Course SOC 2 | 0 | 0
  Undelayed late MTX elimination in Course SOC 2 | 3 | 1
  Delayed late MTX elimination in Course MOD 1 | 0 | 0
  Undelayed late MTX elimination in Course MOD 1 | 2 | 1
  Delayed late MTX elimination in Course MOD 2 | 0 | 1
  Undelayed late MTX elimination in Course MOD 2 | 2 | 0

13. Secondary Outcome: Number of Grade A1, Grade A2, Grade B, Grade C, or Grade D Excretion Toxicities as Listed in the MTX-toxicity Management Instructions
Description: The MTX-toxicity management instructions provided in the protocol are based on the Children's Oncology Group (COG) treatment management recommendations used in study protocol AOST0331, EURAMOS 1. The COG recommend changes in the hydration and the rescue frequency and/or dose to be done if pre-specified toxicities of different severity grades occur.
Time Frame: Time from start of MTX treatment until serum MTX level is ≤ 0.1 μmol/L
Population: The All Patients Treated Set (APTS) included all patients receiving at least one bolus injection of Modufolin (MOD).
Measure: Number; unit: Number of MTX excretion toxicities
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 4 | 4
Number of MTX excretion toxicities
  Grade A2 (24h) SOC 1 | 2 | 2
  Grade A2 (24h) SOC 2 | 2 | 2
  Grade A2 (24h) MOD 1 | 1 | 3
  Grade A2 (24h) MOD 2 | 2 | 1
  Grade B (24h) SOC 1 | 1 | 0
  Grade B (24h) SOC 2 | 0 | 0
  Grade B (24h) MOD 1 | 1 | 0
  Grade B (24h) MOD 2 | 1 | 1
  None (24h) SOC 1 | 1 | 2
  None (24h) SOC 2 | 2 | 2
  None (24h) MOD 1 | 2 | 1
  None (24h) MOD 2 | 1 | 1
  Grade A2 (48h) SOC 1 | 1 | 2
  Grade A2 (48h) SOC 2 | 1 | 1
  Grade A2 (48h) MOD 1 | 2 | 2
  Grade A2 (48h) MOD 2 | 2 | 1
  Grade B (48h) SOC 1 | 1 | 0
  Grade B (48h) SOC 2 | 0 | 0
  Grade B (48h) MOD 1 | 0 | 0
  Grade B (48h) MOD 2 | 0 | 1
  None (48h) SOC 1 | 2 | 2
  None (48h) SOC 2 | 3 | 3
  None (48h) MOD 1 | 2 | 2
  None (48h) MOD 2 | 2 | 1
  Grade A1 (72h) SOC 1 | 2 | 0
  Grade A1 (72h) SOC 2 | 2 | 1
  Grade A1 (72h) MOD 1 | 1 | 1
  Grade A1 (72h) MOD 2 | 2 | 0
  Grade A2 (72h) SOC 1 | 1 | 0
  Grade A2 (72h) SOC 2 | 1 | 0
  Grade A2 (72h) MOD 1 | 1 | 0
  Grade A2 (72h) MOD 2 | 0 | 0
  Grade B (72h) SOC 1 | 0 | 0
  Grade B (72h) SOC 2 | 0 | 0
  Grade B (72h) MOD 1 | 0 | 0
  Grade B (72h) MOD 2 | 0 | 1
  None (72h) SOC 1 | 1 | 4
  None (72h) SOC 2 | 1 | 3
  None (72h) MOD 1 | 2 | 3
  None (72h) MOD 2 | 2 | 2

14. Secondary Outcome: Characterization (Number/Severity) of All Reported AEs During the ENTIRE STUDY PERIOD.
Description: The severity of AEs have been done using NCI CTCAE v4.0. Total number of AEs per severity grade are presented for all AEs and for AEs related to MTX. For AEs related to MTX the number of AEs occurring per preferred term and severity grade are detailed.The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE; Grade 1 Mild, Grade 2 Moderate, Grade 3 Severe, Grade 4 Life-threatening, and Grade 5 Death related to AE.
Time Frame: From the start of HDMTX administration through 8 days post dose for all 4 courses of HDMTX in total
Population: The All Patients Treated Set (APTS) included all patients receiving at least one bolus injection of Modufolin (MOD).
Measure: Number; unit: Number of AEs
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 4 | 4
Number of AEs
  Grade 1 (ALL AEs) | 40 | 27
  Grade 2 (ALL AEs) | 8 | 15
  Grade 3 (ALL AEs) | 11 | 6
  Grade 4 (ALL AEs) | 3 | 9
  Any Grade (ALL AEs) | 62 | 49
  Grade 1 (AEs Related to MTX) | 25 | 20
  Grade 2 (AEs Related to MTX) | 6 | 12
  Grade 3 (AEs Related to MTX) | 6 | 5
  Grade 4 (AEs Related to MTX) | 1 | 1
  Any Grade (AEs Related to MTX) | 38 | 38
  ALAT increase (Related to MTX) Grade 1 | 2 | 0
  ALAT increase (Related to MTX) Grade 2 | 1 | 3
  ALAT increase (Related to MTX) Grade 3 | 4 | 0
  ALAT increase (Related to MTX) Grade 4 | 1 | 0
  ALAT increase (Related to MTX) Any Grade | 8 | 3
  Anemia (Related to MTX) Grade 1 | 3 | 0
  Anemia (Related to MTX) Grade 2 | 4 | 0
  Anemia (Related to MTX) Grade 3 | 0 | 0
  Anemia (Related to MTX) Grade 4 | 0 | 0
  Anemia (Related to MTX) Any Grade | 7 | 0
  ASAT increased (Related to MTX) Grade 1 | 5 | 2
  ASAT increased (Related to MTX) Grade 2 | 0 | 0
  ASAT increased (Related to MTX) Grade 3 | 2 | 0
  ASAT increased (Related to MTX) Grade 4 | 0 | 0
  ASAT increased (Related to MTX) Any Grade | 7 | 2
  Cheilitis (Related to MTX) Grade 1 | 0 | 1
  Cheilitis (Related to MTX) Grade 2 | 0 | 2
  Cheilitis (Related to MTX) Grade 3 | 0 | 0
  Cheilitis (Related to MTX) Grade 4 | 0 | 0
  Cheilitis (Related to MTX) Any Grade | 0 | 0
  Convulsion (Related to MTX) Grade 1 | 0 | 0
  Convulsion (Related to MTX) Grade 2 | 0 | 0
  Convulsion (Related to MTX) Grade 3 | 0 | 1
  Convulsion (Related to MTX) Grade 4 | 0 | 0
  Convulsion (Related to MTX) Any Grade | 0 | 1
  Diarrhoea (Related to MTX) Grade 1 | 2 | 0
  Diarrhoea (Related to MTX) Grade 2 | 1 | 0
  Diarrhoea (Related to MTX) Grade 3 | 0 | 0
  Diarrhoea (Related to MTX) Grade 4 | 0 | 0
  Diarrhoea (Related to MTX) Any Grade | 3 | 0
  Drug clearance decreased (Related to MTX) Grade 1 | 0 | 1
  Drug clearance decreased (Related to MTX) Grade 2 | 0 | 0
  Drug clearance decreased (Related to MTX) Grade 3 | 0 | 0
  Drug clearance decreased (Related to MTX) Grade 4 | 0 | 0
  Drug clearance decreased (Related to MTX) AnyGrade | 0 | 1
  Febrile neutropenia (Related to MTX) Grade 1 | 0 | 0
  Febrile neutropenia (Related to MTX) Grade 2 | 0 | 0
  Febrile neutropenia (Related to MTX) Grade 3 | 0 | 1
  Febrile neutropenia (Related to MTX) Grade 4 | 0 | 0
  Febrile neutropenia (Related to MTX) Any Grade | 0 | 1
  Headache (Related to MTX) Grade 1 | 1 | 0
  Headache (Related to MTX) Grade 2 | 0 | 1
  Headache (Related to MTX) Grade 3 | 0 | 0
  Headache (Related to MTX) Grade 4 | 0 | 0
  Headache (Related to MTX) Any Grade | 1 | 1
  Nausea (Related to MTX) Grade 1 | 2 | 4
  Nausea (Related to MTX) Grade 2 | 0 | 2
  Nausea (Related to MTX) Grade 3 | 0 | 0
  Nausea (Related to MTX) Grade 4 | 0 | 0
  Nausea (Related to MTX) Any Grade | 2 | 6
  Nephropathy (Related to MTX) Grade 1 | 0 | 1
  Nephropathy (Related to MTX) Grade 21 | 0 | 0
  Nephropathy (Related to MTX) Grade 3 | 0 | 0
  Nephropathy (Related to MTX) Grade 4 | 0 | 0
  Nephropathy (Related to MTX) Any Grade | 0 | 1
  Neutropenia (Related to MTX) Grade 1 | 0 | 0
  Neutropenia (Related to MTX) Grade 2 | 0 | 0
  Neutropenia (Related to MTX) Grade 3 | 0 | 0
  Neutropenia (Related to MTX) Grade 4 | 0 | 1
  Neutropenia (Related to MTX) Any Grade | 0 | 1
  Neutrophil count decrease (Related to MTX) Grade 1 | 0 | 0
  Neutrophil count decrease (Related to MTX) Grade 2 | 0 | 0
  Neutrophil count decrease (Related to MTX) Grade 3 | 0 | 1
  Neutrophil count decrease (Related to MTX) Grade 4 | 0 | 0
  Neutrophil count decrease (Related to MTX)AnyGrade | 0 | 1
  Pyrexia (Related to MTX) Grade 1 | 1 | 0
  Pyrexia (Related to MTX) Grade 2 | 0 | 0
  Pyrexia (Related to MTX) Grade 3 | 0 | 0
  Pyrexia (Related to MTX) Grade 4 | 0 | 0
  Pyrexia (Related to MTX) Any Grade | 1 | 0
  Stomatitis (Related to MTX) Grade 1 | 0 | 3
  Stomatitis (Related to MTX) Grade 2 | 0 | 2
  Stomatitis (Related to MTX) Grade 3 | 0 | 1
  Stomatitis (Related to MTX) Grade 4 | 0 | 0
  Stomatitis (Related to MTX) Any Grade | 0 | 6
  Vomiting (Related to MTX) Grade 1 | 9 | 8
  Vomiting (Related to MTX) Grade 2 | 0 | 2
  Vomiting (Related to MTX) Grade 3 | 0 | 0
  Vomiting (Related to MTX) Grade 4 | 0 | 0
  Vomiting (Related to MTX) Any Grade | 9 | 10
  WBC count decreased (Related to MTX) Grade 1 | 0 | 0
  WBC count decreased (Related to MTX) Grade 2 | 0 | 0
  WBC count decreased (Related to MTX) Grade 3 | 0 | 1
  WBC count decreased (Related to MTX) Grade 4 | 0 | 0
  WBC count decreased (Related to MTX) Any Grade | 0 | 1

ADVERSE EVENTS:
Time Frame: 3 years, 1 month
Description: The time-frame for reporting adverse events: From the start of HDMTX administration through 8 days post dose for each course of HDMTX.
Groups:
- Cohort 1: 1 MAP cycle (incl. 2 HDMTX courses with SOC rescue 15mg/m2)
  1 MAP cycle (incl. 2 HDMTX courses with MOD rescue 15mg/m2)
  SOC was administered as rescue in the 2 first HDMTX courses and MOD in the 2 following courses.
  Treatment according to the MAP schedule applied. SOC or MOD commenced 24 h after administration of HDMTX and then every 6 h until the serum-MTX levels were ≤ 0.1 µmol/L, in accordance with COG management recommendations.
- Cohort 2: 1 MAP cycle (incl. 2 HDMTX courses with SOC rescue 15mg/m2)
  1 MAP cycle (incl. 2 HDMTX courses with MOD rescue 7.5mg/m2)
  SOC was administered as rescue in the 2 first HDMTX courses and MOD in the 2 following courses.
  Treatment according to the MAP schedule applied. SOC or MOD commenced 24 h after administration of HDMTX and then every 6 h until the serum-MTX levels were ≤ 0.1 µmol/L, in accordance with COG management recommendations.
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 2/8 | 3/10
Other Adverse Events (participants affected / at risk) | 4/8 | 4/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=8) | Cohort 2 (N=10)
Platelet count decreased (Investigations) | 1 (3) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Candida sepsis (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Cohort 1 (N=8) | Cohort 2 (N=10)
Alanine aminotransferase increased (Investigations) | 2 (8) | 1 (3)
Aspartate aminotransferase increased (Investigations) | 2 (7) | 1 (2)
Drug clearance decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (2) | 1/4 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (9) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 2 (3)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (7)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 2 (4)
Vomiting (Gastrointestinal disorders) | 4 (14) | 4 (13)
Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bacterial disease carrier (Infections and infestations) | 1 (1) | 0 (0)
Cheilitis (Infections and infestations) | 0 (0) | 1 (3)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At least 30 d prior to submission the PI shall provide the Sponsor with results communication for review. The Sponsor shall notify the PI in writing about the review outcome within 30 d from receipt. No public release shall be made unless the Sponsor has consented in writing. The Sponsor may notify the PI that the material shall be withhold from submission for 90 days more to allow filing of applications to secure IPR or to take such measures to establish and preserve its proprietary rights.